CLINICAL TRIAL: NCT00416351
Title: A Phase I/II Study of Clofarabine in Patients With Relapsed T-Cell and NK-Cell Lymphomas
Brief Title: Clofarabine in Treating Patients With T-Cell or Natural Killer-Cell Non-Hodgkin's Lymphoma That Has Relapsed or Not Responded to Previous Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Rochester (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-065; P30CA008748 (NIH); MSKCC-06065
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-03

CONDITIONS: Leukemia; Lymphoma; Small Intestine Cancer
Keywords: anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult nasal type extranodal NK/T-cell lymphoma; prolymphocytic leukemia; childhood nasal type extranodal NK/T-cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Leukemia, Prolymphocytic; Lymphoma, T-Cell, Cutaneous | interventions — Clofarabine

ARMS (1):
- Clofarabine (Experimental): Patients will receive intravenous clofarabine once daily for three consecutive days. Doses of clofarabine will start at 4 mg/m2/day and will be escalated to higher dose levels.
  Interventions: Drug: clofarabine

INTERVENTIONS:
Drug: clofarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I/II trial is studying the side effects and best dose of clofarabine and to see how well it works in treating patients with T-cell or natural killer-cell lymphoma that has relapsed or not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of clofarabine in patients with relapsed or refractory T-cell or natural killer-cell lymphoma.
* Determine the toxicity of this drug in these patients.
* Determine, preliminarily, the efficacy of this drug, in terms of response rate, in these patients.

OUTLINE: This is a phase I, non-randomized, dose-escalation study followed by an open-label, phase II study.

* Phase I: Patients receive clofarabine IV over 1 hour once daily on days 1-3. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or partial response (PR) or complete response (CR) may receive 2 additional courses of treatment. Patients with PR or CR after completing 4 courses of therapy may receive 2 additional courses.

Cohorts of 1-6 patients receive escalating doses of clofarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive clofarabine as in phase I at the MTD determined in phase I.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed T-cell or natural killer (NK)-cell lymphoma, including any of the following subtypes:

  * Blastic NK-cell lymphoma
  * T/NK-cell lymphoma/leukemia
  * Adult T-cell lymphoma/leukemia
  * T-cell prolymphocytic leukemia
  * T-lymphoblastic lymphoma
  * Peripheral T-cell lymphoma, not otherwise specified
  * Angioimmunoblastic T-cell lymphoma
  * Anaplastic large cell lymphoma
  * Transformed mycosis fungoides
  * Subcutaneous panniculitis-like T-cell lymphoma
  * Nasal T/NK-cell lymphoma
  * Enteropathy-type T-cell lymphoma
  * Hepatosplenic gamma/delta T-cell lymphoma
* Relapsed or refractory disease, meeting both of the following criteria:

  * Must have been treated with prior cytotoxic chemotherapy and/or monoclonal antibody therapy
  * No standard curative treatment exists

    * Allogeneic bone marrow transplantation is not considered standard curative treatment
* Evaluable disease (Phase I)
* Measurable disease, defined as any nodal site or mass lesion ≥ 1.5 cm in longest transverse diameter on physical exam or CT scan OR a measurable extranodal site > 1 cm (Phase II)

  * Patients with evaluable blood- or marrow-based disease are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³ (Phase I)
* Absolute neutrophil count ≥ 500/mm³ (Phase II)
* Platelet count ≥ 100,000/mm³ (Phase I)
* Platelet count ≥ 50,000/mm³ (Phase II)
* Creatinine < 2.0 mg/dL*
* Bilirubin ≤ 2.0 times upper limit of normal (ULN)*
* AST and ALT ≤ 2.5 times ULN*
* No active infection requiring antibiotics
* No New York Heart Association class III or IV congestive heart failure
* No known HIV positivity
* No other active malignancy requiring therapy
* No other serious or life-threatening condition deemed unacceptable by the principal investigator
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception NOTE: *Unless due to lymphoma and patients are entering to the phase II portion of the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior therapy, including any of the following:

  * Interferon
  * Antibody therapy
  * Retinoids
  * Other non-chemotherapeutic treatment
* Concurrent stable-dose corticosteroids allowed
* No colony-stimulating factor therapy during the first course of study therapy

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-06-27 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- 4 mg/m2/Day Clofarabine; 8 mg/m2/Day Clofarabine; 13.2 mg/m2/Day Clofarabine; 20 mg/m2/Day Clofarabine; 28 mg/m2/Day Clofarabine: Patients will receive intravenous clofarabine once daily for three consecutive days. Doses of clofarabine will start at 4 mg/m2/day and will be escalated to higher dose levels.
Period: Overall Study
Arm/Group | 4 mg/m2/Day Clofarabine | 8 mg/m2/Day Clofarabine | 13.2 mg/m2/Day Clofarabine | 20 mg/m2/Day Clofarabine | 28 mg/m2/Day Clofarabine
Started | 1 | 3 | 4 | 17 | 4
Completed | 1 | 3 | 4 | 17 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg/m2/Day Clofarabine | 8 mg/m2/Day Clofarabine | 13.2 mg/m2/Day Clofarabine | 20 mg/m2/Day Clofarabine | 28 mg/m2/Day Clofarabine | Total
Number analyzed (Participants) | 1 | 3 | 4 | 17 | 4 | 29
Age, Continuous [Mean (Full Range); unit: years] | 62 [62 to 62] | 65.3 [37 to 80] | 58 [44 to 79] | 54.1 [23 to 76] | 54.5 [35 to 71] | 59 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 9 | 0 | 14
  Male | 0 | 1 | 2 | 8 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 4 | 17 | 4 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 5 | 2 | 7
  White | 0 | 3 | 3 | 10 | 2 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 3 | 4 | 17 | 4 | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Time Frame: 2 years
Measure: Number; unit: mg/m2 of clofarabine
Groups:
- Clofarabine: Patients will receive intravenous clofarabine once daily for three consecutive days. Doses of clofarabine will start at 4 mg/m2/day and will be escalated to higher dose levels.
  clofarabine
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
mg/m2 of clofarabine | 20

2. Primary Outcome: Response Rate for Participants With Non-Hodgkin's Lymphoma
Description: Response rate as defined by complete remission, complete remission unconfirmed, partial remission, positron emission tomography (PET)-negative partial remission, stable disease, and progressive disease (Phase II)
Time Frame: 2 years
Population: Evaluable participants with Non-Hodgkin's Lymphoma
Measure: Count of Participants; unit: Participants
Groups:
- 8 mg/m2/Day Clofarabine: Patients will receive intravenous clofarabine once daily for three consecutive days. Doses of clofarabine will start at 8 mg/m2/day and will be escalated to higher dose levels.
- 13.2 mg/m2/Day Clofarabine: Patients will receive intravenous clofarabine once daily for three consecutive days. Doses of clofarabine will start at 13.2 mg/m2/day and will be escalated to higher dose levels.
- 20 mg/m2/Day Clofarabine: Patients will receive intravenous clofarabine once daily for three consecutive days. Doses of clofarabine will start at 20 mg/m2/day and will be escalated to higher dose levels.
- 28 mg/m2/Day Clofarabine: Patients will receive intravenous clofarabine once daily for three consecutive days. Doses of clofarabine will start at 28 mg/m2/day and will be escalated to higher dose levels.
Arm/Group | 4 mg/m2/Day Clofarabine | 8 mg/m2/Day Clofarabine | 13.2 mg/m2/Day Clofarabine | 20 mg/m2/Day Clofarabine | 28 mg/m2/Day Clofarabine
Number analyzed (Participants) | 1 | 3 | 4 | 17 | 4
Participants
  Complete Response | 0 | 1 | 1 | 1 | 0
  Partial Response (PR) | 0 | 0 | 0 | 1 | 0
  Stable Disease (SD) | 0 | 1 | 0 | 2 | 1
  Progression of Disease (POD) | 1 | 1 | 2 | 11 | 3
  Not Evaluable | 0 | 0 | 0 | 0 | 0
  Stable Disease/Progression of Disease (SD/POD) | 0 | 0 | 1 | 2 | 0

3. Secondary Outcome: Participants Evaluated for Toxicity
Description: Toxicity as defined by NCI Common Terminology Criteria for Adverse Events v 3.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg/m2/Day Clofarabine | 8 mg/m2/Day Clofarabine | 13.2 mg/m2/Day Clofarabine | 20 mg/m2/Day Clofarabine | 28 mg/m2/Day Clofarabine
Number analyzed (Participants) | 1 | 3 | 4 | 17 | 4
Participants | 1 | 3 | 4 | 17 | 4

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 4 mg/m2/Day Clofarabine | 8 mg/m2/Day Clofarabine | 13.2 mg/m2/Day Clofarabine | 20 mg/m2/Day Clofarabine | 28 mg/m2/Day Clofarabine
All-Cause Mortality (participants affected / at risk) | 1/1 | 3/3 | 3/4 | 12/17 | 4/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 1/4 | 13/17 | 4/4
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 4/4 | 17/17 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg/m2/Day Clofarabine (N=1) | 8 mg/m2/Day Clofarabine (N=3) | 13.2 mg/m2/Day Clofarabine (N=4) | 20 mg/m2/Day Clofarabine (N=17) | 28 mg/m2/Day Clofarabine (N=4)
Calcium, high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Creatinine (Investigations) | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1
Fever (in the absence of neutropenia) (General disorders) | 0 | 0 | 0 | 2 | 0
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Inf norm ANC/gr1/2 neut-Bronchitis NOS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Inf norm ANC/gr1/2 neut-Joint (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Inf unknown ANC-Cellulitis(skin) (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Inf unknown ANC-Pneumonia(lung) (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection w/ Gr 3/4 neut, Blood (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection, other (Infections and infestations) | 0 | 0 | 0 | 6 | 0
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 0 | 0 | 1 | 0
Ocular/Visual - Other (specify) (Eye disorders) | 0 | 0 | 0 | 1 | 0
Odor (patient odor) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain - Other (specify) (General disorders) | 0 | 0 | 0 | 2 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Platelets (Investigations) | 0 | 0 | 0 | 2 | 0
Pleural effusion (non-malig) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rigors/chills (General disorders) | 0 | 0 | 0 | 0 | 1
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Uric acid, high (hyperuricemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg/m2/Day Clofarabine (N=1) | 8 mg/m2/Day Clofarabine (N=3) | 13.2 mg/m2/Day Clofarabine (N=4) | 20 mg/m2/Day Clofarabine (N=17) | 28 mg/m2/Day Clofarabine (N=4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 2 | 2 | 2 | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Hemoglobin (Investigations) | 0 | 2 | 1 | 10 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pain - Other (specify) (General disorders) | 0 | 0 | 1 | 1 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (General disorders) | 0 | 1 | 0 | 0 | 1
Creatinine (Investigations) | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Infection, other (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Leukocytes (total WBC) (Investigations) | 0 | 3 | 2 | 10 | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 3 | 2 | 9 | 3
Pain - Oral cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Platelets (Investigations) | 0 | 2 | 2 | 10 | 4
Pleural effusion (non-malig) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
ALT, SGPT (Investigations) | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
AST, SGOT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 0 | 1 | 1 | 0
Calcium, high (hypercalcemia) (Investigations) | 0 | 0 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Edema: Limb (General disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1
Infection w/ Gr 3/4 neut, Skin (cellulites) (Infections and infestations) | 0 | 0 | 0 | 1 | 0
INR (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphopenia (Investigations) | 1 | 2 | 2 | 11 | 3
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 | 0 | 0 | 1 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 1
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Rigors/chills (General disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-08-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT00416351/Prot_SAP_000.pdf